CLINICAL TRIAL: NCT03421977
Title: A Long Term Follow up Safety Study of Patients in the AVXS-101-CL-101 Gene Replacement Therapy Clinical Trial for Spinal Muscular Atrophy Type 1 Delivering AVXS 101
Brief Title: Long-Term Follow-up Study for Patients From AVXS-101-CL-101
Acronym: START
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: AVXS-101-LT-001; COAV101A12401 (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Spinal Muscular Atrophy 1
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — Zolgensma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: Onasemnogene Abeparvovec-xioi — Patients received treatment with onasemnogene abeparvovec-xioi in the parent study, AVXS-101-CL-101
  Other Names: Zolgensma

SUMMARY:
This is a long term, safety follow up study of patients in the AVXS-101-CL-101 gene replacement therapy clinical trial for SMA Type 1 delivering onasemnogene abeparvovec-xioi. Patients will roll over from the parent study into this long-term study for continuous safety monitoring for up to 15 years.

DETAILED DESCRIPTION:
This is a long term, safety follow up study of patients in the AVXS-101-CL-101 gene replacement therapy clinical trial for SMA Type 1 delivering onasemnogene abeparvovec-xioi. Patients will roll over from the parent study into this long-term study for continuous safety monitoring for up to 15 years. The last visit of the parent study or early discontinuation from the parent study may serve as the visit at which the informed consent form process is conducted for the AVXS 101-LT-001 long term follow-up safety study. Patients will return annually for follow up study visits for five (5) years, and then will be contacted via phone annually for ten (10) years. Additionally, patient record transfers from their local physician and/or neurologist will be requested in conjunction with the annual study visits and phone contacts for review by the investigator.

If the patient is unable to return to the original investigative site, the sponsor will arrange with the patients' local established physician to serve as an additional investigator to conduct the required assessments.

This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Inclusion Criteria:

1. Patient who received onasemnogene abeparvovec-xioi in the AVXS-101-CL-101 gene replacement therapy clinical trial for SMA Type 1.
2. Parent/legal guardian willing and able to complete the informed consent process, comply with study procedures and visit schedule.

Exclusion Criteria:

1. Parent/legal guardian unable or unwilling to participate in the long term follow up safety study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the AVXS-101-CL-101 gene replacement therapy clinical trial for SMA Type 1 delivering onasemnogene abeparvovec-xioi will roll over from the previous study into the AVXS-101-LT-001 study for continuous safety monitoring for up to 15 years.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2030-12-02 (Estimated); Study Completion 2030-12-02 (Estimated)

PRIMARY OUTCOMES:
Long-Term Safety | 15 years
  The primary objective is to collect long term safety data of patients with SMA Type 1 who were treated with onasemnogene abeparvovec-xioi in the AVXS-101-CL-101 gene replacement therapy clinical trial by assessing incidence of SAEs and Adverse Events of Special Interest

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Day JW, Mendell JR, Mercuri E, Finkel RS, Strauss KA, Kleyn A, Tauscher-Wisniewski S, Tukov FF, Reyna SP, Chand DH. Clinical Trial and Postmarketing Safety of Onasemnogene Abeparvovec Therapy. Drug Saf. 2021 Oct;44(10):1109-1119. doi: 10.1007/s40264-021-01107-6. Epub 2021 Aug 12. PMID 34383289
- [Derived] Mendell JR, Al-Zaidy SA, Lehman KJ, McColly M, Lowes LP, Alfano LN, Reash NF, Iammarino MA, Church KR, Kleyn A, Meriggioli MN, Shell R. Five-Year Extension Results of the Phase 1 START Trial of Onasemnogene Abeparvovec in Spinal Muscular Atrophy. JAMA Neurol. 2021 Jul 1;78(7):834-841. doi: 10.1001/jamaneurol.2021.1272. PMID 33999158